CLINICAL TRIAL: NCT04581486
Title: Evaluation of the Effectiveness of an Optimal-Massive Intervention in Older Patients With Oropharyngeal Dysphagia
Brief Title: Effectiveness of an Optimal-Massive Intervention in Older Patients With Dysphagia
Acronym: OMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Mataró (Other)
Collaborators: Nutricia Research (Industry)
Responsible Party: Principal Investigator, Pere Clave, Director of Research and Academic Development at CSdM, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OMI
Record Dates: First submitted 2020-09-15; First posted 2020-10-09 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Swallowing Disorder; Oropharyngeal Dysphagia; Respiratory Infection; Malnutrition; Dehydration; Oral Disease
MeSH Terms: conditions — Deglutition Disorders; Respiratory Tract Infections; Malnutrition; Dehydration; Mouth Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMI intervention (Experimental): Multimodal intervention based on optimal fluid viscosity adaptation (with Nutilis Clear®), optimal nutritional support with a triple adaptation of food (texture, (Nutilis Clear®)) caloric and protein content, organoleptic) + ONS depending on nutritional status and evaluation and optimal treatment of oral hygiene (tooth brushing + antiseptic mouthwash + professional dental cleaning)
  Interventions: Other: Optimal-Massive Intervention
- Control intervention (standard clinical practice) (Other): Standard clinical practice (fluid adaptation with Nutilis Powder® and simple texture adaptation (for solids (Nutilis Powder®))
  Interventions: Other: Control (standard clinical practice)

INTERVENTIONS:
Other: Optimal-Massive Intervention — Multimodal intervention based on 3 main measures: a) optimal fluid viscosity adaptation (with Nutilis Clear®), b) optimal nutritional support with a triple adaptation of food (texture, (Nutilis Clear®)) caloric and protein content, organoleptic) + ONS depending on nutritional status and evaluation and c) optimal treatment of oral hygiene (tooth brushing + antiseptic mouthwash + professional dental cleaning).
  Arms: OMI intervention
Other: Control (standard clinical practice) — Standard clinical practice (fluid adaptation with Nutilis Powder® and simple texture adaptation (for solids (Nutilis Powder®))
  Arms: Control intervention (standard clinical practice)

SUMMARY:
The aim of this study is to evaluate the efficacy of an optimal-massive intervention (OMI) based on increasing shear viscosity of fluids, nutritional support with oral nutritional supplements (ONS) and triple adaptation of food (rheological and textural, caloric and protein and organoleptic) and oral hygiene improvement on the incidence of respiratory infections in older patients with OD. We have designed a randomized clinical trial, with two parallel arms and 6 months follow-up. The study population will be constituted by older patients of 70 years or more with OD hospitalized at Hospital de Mataró by an acute process that will be identified by using the volume-viscosity swallow clinical test. We will consecutively recruit 500 subjects during admission (Geriatrics, Internal medicine, etc.) at the Hospital de Mataró. Patients included will be randomly assigned to one of both interventional groups: a) study intervention: multifactorial intervention based on fluid viscosity adaptation (with a xanthan gum thickener -> Nutilis Clear®), nutritional support with a triple adaptation of food (texture, caloric and protein content, organoleptic) + pre-thickened ONS and evaluation and treatment of oral hygiene (tooth brushing + antiseptic mouthwashes + professional dental cleaning), or b) control intervention: standard clinical practice (fluid adaptation with Nutilis Powder and simple texture adaptation for solids). Main outcome measures: respiratory infection incidence during the 6-month period follow-up. Secondary outcomes: mortality at 6 months, general hospital readmissions and readmissions due to respiratory infections, nutritional status, hydration status, quality of life, functional status, oral hygiene and dysphagia severity and its relationship with other study variables.

DETAILED DESCRIPTION:
DESIGN

- Study design: Randomized controlled clinical trial with two parallel arms and 6 months follow-up.

AIMS

* Primary aim: To evaluate the effect of a rheological, nutritional and oral hygiene intervention (OMI) on the incidence of respiratory infections including lower respiratory tract infections -LRTI-, pneumonia and chronic obstructive pulmonary disease (COPD) infectious exacerbations in older patients with OD at 6 months follow-up.
* Secondary aims: to evaluate the effect at 1, 3 and 6 months of this intervention on:

  1. Mortality.
  2. General hospital readmission and hospital readmission due to respiratory infections.
  3. Nutritional status according to the MNA, anthropometrical measures and biochemical markers.
  4. Hydration status according to bioimpedance.
  5. Quality of life according to the EQ-5D.
  6. Functional status according to Barthel index.
  7. Oral hygiene status according to the simplified oral hygiene index (OHI-S).

Other aims:

- To evaluate the effect at 1, 3 and 6 months of this intervention on:

1. Swallowing function according to the V-VST.
2. Rate of institutionalization.
3. Compliance with the treatments (thickeners, ONS, diets and oral health).
4. Palatability and acceptability of diets.
5. To evaluate the relationship between severity of dysphagia (V-VST / FOIS), nutritional status, oral hygiene and the incidence of respiratory infections (LRTI, pneumonia and/or COPD exacerbations).

   STUDY POPULATION

   - Study subjects: 500 older patients with OD admitted to Hospital de Mataró for acute conditions (internal medicine, cardiology, pneumology, neurology, geriatric wards, etc). Number of subjects necessary: 500 (G1: 250; G2: 250): Accepting an α risk of 0.05 and a β risk of 0.2 in a bilateral contrast, 244 subjects in each group are required to detect as statistically significant difference in the percentage of patients with LRTI at six months that for the control group is expected to be 20 % and for the intervention group of 10% (reduction by half).A tracking loss rate of 20% has been assumed and the required number of subjects (244) in each group already includes the dropout rate. Investigators will intend to recruit a total sample of 500* individuals, 250 in each intervention branch.

   SAFETY - Safety and tolerance parameters: Incidence, frequency, seriousness, severity and relatedness of adverse events or serious adverse events.

   STUDY GROUPS AND INTERVENTION

   - Study groups: there will be 2 groups of patients: G1 - study intervention, 250 patients; G2 - control intervention, 250 patients.

   - Study interventions:there will be 2 interventions: G1) study intervention: multimodal intervention based on optimal fluid viscosity adaptation (with Nutilis Clear®), optimal nutritional support with a triple adaptation of food (texture, (Nutilis Clear®)) caloric and protein content, organoleptic) + ONS depending on nutritional status and evaluation and optimal treatment of oral hygiene (tooth brushing + antiseptic mouthwash + professional dental cleaning); G2) control intervention: standard clinical practice (fluid adaptation with Nutilis Powder® and simple texture adaptation (for solids (Nutilis Powder®)).

   STATISTICAL ANALYSIS

   - Statistical analysis: the primary outcome will be the occurrence of the respiratory infections during the follow-up period (number of events/100 patients-year) and will be mainly analyzed with the Poisson regression.

   Qualitative data will be presented as relative and absolute frequencies and analyzed by the Fisher's exact test or the Chi-square test. Volume and viscosity levels (V-VST) will be compared between them by applying the McNemar's test. Continuous data will be presented as mean±standard deviation (SD) and compared with the T-test (intergroup comparisons) or Paired T-test (intragroup comparisons). For those variables that will not follow a normal distribution, the nonparametric Mann-Whitney U-test (intergroup comparisons), the Wilcoxon-paired test (intragroup comparisons) or the Kruskal-Wallis' test for multiple comparisons with Dunn's multiple comparison test will be used. Survival curves will be used to evaluate 6-month mortality after discharge. The primary analysis will be performed on the ITT population. Note: primary analysis is on number of events at 6 months follow-up, to simplify sample size considerations are based on percentage of patients with LRTI at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 70 years or older.
2. Diagnosed oropharyngeal dysphagia (signs of impaired efficacy and/or safety of swallow assessed with the V-VST).
3. Giving written informed consent. In case of dementia or incapacitation, given consent by the nearest relative, main caregiver or legal representative.

Exclusion Criteria:

1. Impaired safety of swallow with 5mL at high viscosity (800 mPa•s for NC).
2. Severe dementia (Pfeiffer >6).
3. Life expectancy less than 6 months.
4. High functional dependence (Barthel index <40, preadmission).
5. Dysphagia caused by anatomical alterations or by head and neck cancer or its treatment.
6. Patients going to nursing home or long-term care at discharge.
7. Participation in any other studies involving investigational or marketed products within four weeks prior to start of the study.
8. Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements.
9. Patients with symptoms suggestive of COVID-19 or confirmed COVID-19.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-06-06 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Respiratory infections incidence. | From discharge to 6 months follow-up
  Respiratory infections incidence (includes LRTI, pneumonia and exacerbations of COPD): all new episodes of respiratory infections recorded in the clinical history or in the reports presented by the patient will be recorded. LRTI: presence of at least 2 of the following symptoms without other cause to explain them: fever, cough, purulent expectoration, rhonchi or wheezing. Pneumonia: performing 1 or more radiographic tests with new condensation, fever or leukopenia or leukocytosis and at least: cough, purulent expectoration, dyspnea, tachypnea, suggestive auscultation or worsening of gas exchange. COPD exacerbation: acute exacerbation of COPD is a sudden worsening of COPD symptoms (shortness of breath, quantity and color of phlegm) that typically lasts for several days. It may be triggered by an infection with bacteria or viruses or by environmental pollutants.

SECONDARY OUTCOMES:
Mortality | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Mortality: the date and reason for death will be recorded (hospitalization, 1, 3 and 6 months).
General readmissions and readmissions for respiratory infections | Through study completion, at 1, 3 and 6 months from disharge.
  General readmissions and readmissions for respiratory infections (1, 3 and 6 months): LRTI, pneumonia and exacerbations of COPD: the reason for admission will be that stated in the hospital database (CMBDAH) according to CIM-10. The information source of the readmissions will be the registration of hospital discharges that is integrated into the hospital information system and that includes the CIM-10 codes of the main and secondary diagnoses of the episode that caused the admission, the date of admission and discharge and the days of hospitalization. Readmissions from pneumonia (codes CIM-10): J13, J18.1, J15.1, J14, J15.4, J15.211, J15.5, A48.1, J15.8, J18.0, J18.8, J69.0; readmissions for LRTI (no pneumonic): J20.0 - J20.9, J10.1, J11.1, J41.8, J44.1 and J44.0. Readmissions from exacerbation of COPD: J441.
Nutritional status (MNA) | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Mini-nutritional assessment form (MNA) (hospitalization, 1, 3 and 6 months).
Nutritional status (Anthropometric measures) | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Heigh in cm (hospitalization, 1, 3 and 6 months).
Nutritional status (Anthropometric measures2) | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Weight in kg (hospitalization, 1, 3 and 6 months).
Nutritional status (Biochemical parameters) | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Biochemical parameters from blood analysis (hospitalization, 3 and 6 months).
Hydration status (bioimpedance) | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Hydration status: we will register total body water and intracellular water with bioimpedance (hospitalization, 1, 3 and 6 months).
Quality of life of patients during the study period | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Quality of life: EQ-5D questionnaire will be used (hospitalization, 1, 3 and 6 months).
Functional status | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Functional status: we will use the Barthel Index (hospitalization, 1, 3 and 6 months).
Oral Hygiene | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Oral Hygiene: the OHI-S (simplified oroal hygiene index) will be collected (hospitalization, 1, 3 and 6 months).
Dysphagia severity | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Severity of dysphagia: according to the different viscosities that patients will be able to swallow and with the Functional Oral Intake Scale (V-VST/FOIS) (hospitalization, 1, 3 and 6 months).

OTHER OUTCOMES:
Sociodemographics | Baseline
  Sociodemographic characteristics of the study population.
Swallowing function (V-VST) | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Swallowing function (V-VST) (hospitalization, 1, 3 and 6 months).
Institutionalization | Through study completion, at 1, 3 and 6 months from disharge.
  Rate of institutionalization (1, 3 and 6 months).
Pharmacological treatment | Baseline
  Drugs taken by the patient.
Geriatric syndromes | Baseline
  Geriatric syndromes
Frailty 1 | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Fried criteria (hospitalization, 1, 3 and 6 months).
Frailty 2 | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Edmonton frail scale (hospitalization, 1, 3 and 6 months).
Toxic habits | Baseline
  Smoking and alcohol consumption
Compliance | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Compliance with the recommendations of the study intervention (adaptations of fluid, prescribed diets and oral hygiene) (hospitalization, 1, 3 and 6 months).
Palatability | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Palatability of the intervention products will be measured with the 5-point facial hedonic scale (hospitalization, 1, 3 and 6 months).
Acceptability | Through study completion, during hospitalization, and at 1, 3 and 6 months from disharge.
  Acceptability of the dietes will be measured with the Food Action Rating Scale (hospitalization, 1, 3 and 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Pere Clavé, MD, PhD, Principal Investigator — Director of Research and Academic Development at CSdM
Locations (1):
- Consorci Sanitari del Maresme (Hospital de Mataró), Mataró, Barcelona, Spain

REFERENCES:
- [Result] Martin A, Ortega O, Roca M, Arus M, Clave P. Effect of A Minimal-Massive Intervention in Hospitalized Older Patients with Oropharyngeal Dysphagia: A Proof of Concept Study. J Nutr Health Aging. 2018;22(6):739-747. doi: 10.1007/s12603-018-1043-3. PMID 29806864
- [Result] Ortega O, Martin A, Clave P. Diagnosis and Management of Oropharyngeal Dysphagia Among Older Persons, State of the Art. J Am Med Dir Assoc. 2017 Jul 1;18(7):576-582. doi: 10.1016/j.jamda.2017.02.015. Epub 2017 Apr 12. PMID 28412164